CLINICAL TRIAL: NCT05399589
Title: Clinical Efficacy of Nobel Parallel CC Implants With on1 Abutment in Posterior Area Participants Participants: Fuming He, Jimin Jiang, Hongye Lu To Evaluate the Long-term Efficacy of on1 Abutment Produced by Nobel Biocare Manufacturer
Brief Title: Clinical Efficacy of Nobel Parallel CC Implants With on1 Abutment in Posterior Area Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DHZhejiangU - 2022(33)
Record Dates: First submitted 2022-05-02; First posted 2022-06-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Failure of Dental Implant Nos
Keywords: Dental implants; One abutment one time; Submerged healing; Bone Remodeling; Definitive abutment
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- on1 abutment (Experimental): The on1 abutment was directly used in the operation to protect the soft tissue mucosa. After three months, the mold was taken directly for formal teeth.
  Interventions: Combination Product: use on1 abutment instead of healing cap in test group
- healing cap (Active Comparator): After the operation, the embedded healing is selected. After waiting for three months, the second stage operation is needed to expose the healing cap
  Interventions: Combination Product: use healing cap in control group

INTERVENTIONS:
Combination Product: use on1 abutment instead of healing cap in test group — We will use on1 abutment instead of healing cap in a implant operation, since the former can protect the soft tissue barrier to a certain extent.
  Arms: on1 abutment
Combination Product: use healing cap in control group — use healing cap in control group
  Arms: healing cap

SUMMARY:
1. Research background NobelBiocare manufacture put forward a new abutment called on1. This concept is based on a two-stage abutment in which the on1 abutment is placed directly on the implant during surgery and will not be disconnected since then. At present, there are very a few clinical prospective studies about clinical effect of Nobelparallel CC implant combined with on1 abutment.
2. Research objective This study will evaluate the clinical efficacy of Nobel parallel with on1 abutment compared to traditional healing cap in posterior teeth in a short term(one year) and long trem (five year) follow-up.
3. Study design and methods:

Design type: prospective clinical study. Study duration: 5 years Start time: From the date of adoption of ethics. End time: 2026. Follow up examination: Panoramic images will be taken at all times to measure the marginal bone level of the implant. Clinical examination and questionnaire survey will be conducted to obtain the implant conditions and patients' satisfaction. Periodontal indexes such as keratinized gingival width, plaque index, gingival index, bleeding on probe, probing depth of peri-implant tissue will be evaluate.

DETAILED DESCRIPTION:
1. Research background NobelBiocare manufacture put forward a new abutment called on1. This concept is based on a two-stage abutment in which the on1 abutment is placed directly on the implant during surgery and will not be disconnected since then. At present, there are very a few clinical prospective studies about clinical effect of Nobelparallel CC implant combined with on1 abutment.
2. Research objective This study will evaluate the clinical efficacy of Nobel parallel with on1 abutment compared to traditional healing cap in posterior teeth during a five-year follow-up.
3. Study design and methods:

Design type: prospective clinical study (Non randomized clinical trial) Study duration: 5 years Start time: From the date of adoption of ethics. End time: 2026. Follow up examination: Panoramic images will be taken at all times to measure the marginal bone level of the implant. Clinical examination and questionnaire survey will be conducted to obtain the implant conditions and patients' satisfaction. Periodontal indexes such as keratinized gingival width, plaque index, gingival index, bleeding on probe, probing depth of peri-implant tissue will be evaluate.

Introduction to the research scheme: Implants of Nobel Parallel CC will be implanted into the posterior teeth in the Affiliated Stomatology Hospital, Zhejiang University School of Medicine since the date of ethical adoption. Forty patients with on1 abutment will be placed with implant. Forty patients with common healing abutment will be selected with the same implants simultaneously. Panoramic images will be evaluated before surgery, immediately after surgery, immediately, 3 months, 1 year, 2 years, 3 years and 4 years after prosthesis loading. Clinical examination and questionnaire survey will be carried out 4 years after prosthesis loading to obtain periodontal indexes about peri-implant tissues. Through the evaluation of the above experimental data, on1 abutment with implant will be analyzed about the clinical efficacy.

ELIGIBILITY:
The inclusion criteria were as follows:

1. At least eighteen years old without any medical contraindications, able to tolerate dental implant surgery;
2. Planned to implant with Nobel Parallel CC™ in the maxillary or mandible posterior tooth regions with single-implant-prosthesis design;
3. No requirement for further bone augmentation;
4. Sufficient space to place the abutment and future prosthesis;
5. Adhere to follow-up.

The exclusion criteria were as follows:

1. Uncontrolled systematic diseases (blood pressure >180/100 mmHg, fasting blood glucose >8.88 mmol/L, myocardial infarction in six months, cardiac function class III to IV, third- or second-degree II atrioventricular block, and double bundle branch block et al.);
2. Using drugs such as bisphosphonates within three months;
3. Heavy smoker (≥ 10 cigarettes per day), alcoholism, and drug abuse;
4. Uncontrolled periodontitis;
5. Implant site infection;
6. Pregnancy or lactation;
7. Severe malocclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
marginal bone level (MBL) | 5 years
  The MBL of the mesial and distal sites of the implants will be measured using panoramic radiograph for the two groups of each period and converted.

CONTACTS AND LOCATIONS:
Overall Officials: Hongye Lu, PhD, Study Chair — this hospital
Locations (1):
- The Affiliated Stomatology Hospital, Zhejiang University School of Medicine, 166 North Qiu'tao Road, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT05399589/Prot_SAP_ICF_000.pdf